CLINICAL TRIAL: NCT04399967
Title: Building Capacity and Promoting Smoking Cessation in the Community Via "Quit to Win" Contest 2020: a Single-blind Randomized Controlled Trial on COVID-19 Related Brief Advice and Personalized Chat-based Intervention for Smoking Cessation
Brief Title: COVID-19 Brief Advice and Chat-based Support for Smoking Cessation Via "Quit to Win" Contest 2020
Acronym: QTW2020
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Council on Smoking and Health (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: QTW 2020
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Quit to Win; COVID-19
MeSH Terms: conditions — Smoking Cessation; COVID-19 | interventions — corticosteroid hormone-induced factor; Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Chat-based support+ COVID-19 specific advice + AWARD advice + COVID-related health warning leaflet + referral card + COSH booklet
  Interventions: Behavioral: Chat-based support; Behavioral: AWARD plus COVID-specific advice; Behavioral: COVID-19 related health warning leaflet; Behavioral: Referral card; Behavioral: COSH Self-help smoking cessation booklet
- Control Group (Experimental): Text-based support + AWARD advice + warning leaflet + referral card + COSH booklet
  Interventions: Behavioral: AWARD advice; Behavioral: Health warning leaflet; Behavioral: SMS-based support; Behavioral: Referral card; Behavioral: COSH Self-help smoking cessation booklet

INTERVENTIONS:
Behavioral: Chat-based support — Participants will receive three months of chat-based support through IM apps (e.g. WhatsApp, WeChat). The regular messages and instant messaging on psychosocial support aim to provide hygienic advice to reduce the risk of exposure to SARS-cov2, increase self-efficacy and confidence, and social support and behavioral capacity of quitting.
  Arms: Intervention Group
Behavioral: AWARD plus COVID-specific advice — Ask about smoking history, Warn about the risks associated with the COVID-19 and smoking (with a COVID-related health warning leaflet), Advise to quit as soon as possible during the COVID-19 pandemic, Refer smokers to SC services (with a referral card, see below for information), and Do it again: to repeat the intervention
  Other Names: Ask, Warn, Advise, Refer, Do-it-again
  Arms: Intervention Group
Behavioral: AWARD advice — Ask about smoking history, Warn about the high risk of smoking, Advise to quit as soon as possible, Refer to the smoking cessation services, and Do it again (if the smokers refused to set quit date).
  Other Names: Ask, Warn, Advise, Refer, Do-it-again
  Arms: Control Group
Behavioral: COVID-19 related health warning leaflet — The 2-sided color printed A4 leaflet, which covers the risk of COVID-19 and smoking and the most important messages to motivate smoking cessation
  Arms: Intervention Group
Behavioral: Health warning leaflet — The 2-sided color printed A4 leaflet, which systematically covers the most important messages to motivate smoking cessation.
  Other Names: Brief leaflet on health warning and smoking cessation
  Arms: Control Group
Behavioral: SMS-based support — Participants will receive regular SMS with similar frequency to Intervention group but with generic information on smoking cessation.
  Arms: Control Group
Behavioral: Referral card — The 3-folded "Smoking Cessation Services" card consists of brief information and highlights of existing smoking cessation services, contact methods, motivation information and strong supporting messages or slogans.
  Other Names: Smoking Cessation Service Card
Behavioral: COSH Self-help smoking cessation booklet — A general smoking cessation self-help booklet

SUMMARY:
The present study will examine (1) the effectiveness of a combined brief advice and personalized chat-based support on COVID-19 related smoking messages and (2) explore the use of CBPR model to build capacity and to engage community partners in taking on this important public health issue for sustainability in the community. In addition, a process evaluation will be conducted to assess the effectiveness of the recruitment activity and how it is linked with the overall program outcomes.

DETAILED DESCRIPTION:
Smoking is detrimental to the immune system and can cause respiratory tract infection. Growing evidence has suggested that compared to non-smokers, COVID-19 patients who have a history of smoking are at a higher risk of developing severe respiratory and cardiovascular symptoms, consequently may require mechanical ventilation and intensive care. A case series of 1,099 COVID-19 patients in China has found that ever smokers, compared with never smokers, were more likely to have severe COVID-19 disease upon hospital admission and be admitted to intensive care unit, need to use mechanical ventilation, and die. The result is corroborated by a multivariable analysis of 78 COVID-19 pneumonia cases in China, which identified smoking as the only preventable risk factor for disease progression. While the link between smoking and the COVID-19 needs further research, smokers appear to be at a greater risk of suffering from serious symptoms due to COVID-19.

The practice of smoking might also predispose smokers to COVID-19 infection. Smoking behavior is characterized by inhalation and the hand-to-mouth movements which increase the possibility of transmission of virus from contaminated fingers and cigarettes to mouth. In Hong Kong, where smoking is banned in indoor public areas and workplace, smokers often gather and smoke at smoking hotspots outdoor, where ashtrays are available. This increases their risk of infection since the smokers are in close contact with each other and have to remove their mask to smoke. Exhaling smoke also aids the spreading the virus in the air. However, misleading information that smoking can prevent COVID-19 infection is widespread on social media.

Public health strategies (e.g., social distancing, staying at home and working from home) may motivate some smokers to reduce or to quit smoking due to the inconvenience to smoke indoor and to buy cigarettes from retail outlets. However, home confinement may result in social isolation and psychological distress (anxiety and stress) both increasing the need for smoking. Some smokers who are not used to smoke at home might be prompted to smoke at home to cope with their craving during lockdown or work from home, which may also expose their family members from second-hand smoke.

Our RCT in QTW Contest 2017 evaluated the effectiveness of a chat-based intervention delivered through a mobile instant messaging application (WhatsApp) plus active referral to SC services to increase quitting. Chat-based intervention resulted in higher abstinence rate compared with the control group at 6-month follow-up. In QTW Contest 2019, we evaluated the effectiveness of a combined intervention of AWARD advice, active referral, instant messaging and optional cocktail intervention to increase abstinence. The preliminary result showed that the personalized instant messaging (PIM) group and regular instant messaging (RIM) group had similar abstinence rate at 6-month follow-up.

Therefore, the present study will examine (1) the effectiveness of a combined brief advice and personalized chat-based support on COVID-19 related smoking messages and (2) explore the use of CBPR model to build capacity and to engage community partners in taking on this important public health issue for sustainability in the community. In addition, a process evaluation will be conducted to assess the effectiveness of the recruitment activity and how it is linked with the overall program outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Smoke at least 1 tobacco stick per day or use e-cigarette daily in the past 3-month
* Able to communicate in Cantonese (including reading Chinese)
* Saliva cotinine 30 ng/ml or above
* Intent to quit / reduce smoking
* Able to use instant messaging tool (e.g., WhatsApp, WeChat) for communication.

Exclusion Criteria:

* Smokers who have communication barrier (either physically or cognitively)
* Smokers who are currently participating in other SC programmes or services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1166 (Actual)
Dates: Start 2020-06-13 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Biochemical validated quit rate | 3-month follow-up
  The primary outcomes are biochemically validated quit rates (exhaled CO < 4 ppm or salivary cotinine < 30 ng/ml) at 3-month in the two groups
Biochemical validated quit rate | 6-month follow-up
  The primary outcomes are biochemically validated quit rates (exhaled CO < 4 ppm or salivary cotinine < 30 ng/ml) at 6-month in the two groups

SECONDARY OUTCOMES:
Smoking quit rate change from baseline at 3-month follow-up | 3-month follow-up
  Self-reported 7-day point prevalence (pp) quit rate at 3-month between the two groups
Smoking quit rate change from baseline at 6-month follow-up | 6-month follow-up
  Self-reported 7-day point prevalence (pp) quit rate at 6-month between the two groups
Smoking reduction rate change from baseline at 3-month follow-up | 3-month follow-up
  Rate of smoking reduction by at least half of baseline amount in the two groups
Smoking reduction rate change from baseline at 6-month follow-up | 6-month follow-up
  Rate of smoking reduction by at least half of baseline amount in the two groups
Engagement in chat-based/text-based support | 3 and 6 months follow-up
  Self-reported engagement in chat-based/SMS-based support in the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Kelvin Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Hong Kong Council on Smoking and Health (COSH), Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weng X, Luk TT, Wu YS, Zhao SZ, Cheung DYT, Tong HSC, Lai VWY, Lam TH, Wang MP. Effect of smoking-related COVID-19 risk messaging on smoking cessation in community smokers: A pragmatic randomized controlled trial. Tob Induc Dis. 2023 Jun 14;21:77. doi: 10.18332/tid/163176. eCollection 2023. PMID 37323509